CLINICAL TRIAL: NCT04406116
Title: Clinical Evaluation of the Safety and Performance of Microwave Coagulation Using the HS1 Instrument for Actual or Potential Non-variceal Bleeding in the Upper Gastrointestinal (GI) Tract
Brief Title: Clinical Evaluation of the Safety and Performance of Microwave Coagulation Using the HS1 Instrument
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Creo Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-HS1-031PRO
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Actual or Potential Nonvariceal Bleeding in the Upper Gastrointestinal (GI) Tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients receiving microwave therapy using the HS1 Instrument (Experimental)
  Interventions: Device: Microwave coagulation using HS1 Instrument

INTERVENTIONS:
Device: Microwave coagulation using HS1 Instrument — Microwave therapy at 5.8 GHz

SUMMARY:
Clinical evaluation of the safety and performance of microwave coagulation using the HS1 Instrument for actual or potential non-variceal bleeding in the upper Gastrointestinal (GI) tract

ELIGIBILITY:
Inclusion Criteria:

* Patient or authorised representative able to comprehend and sign the Informed Consent form.
* Actual or potential non-variceal bleeding in the upper GI, including angiodysplasia or AVM malformations such as Dieulafoy's lesion with a Glasgow-Blatchford score of greater than 1

Exclusion Criteria:

* As stated in the contraindications in the HS1 IFU;
* Aged <18 years of age
* Those described as vulnerable populations in EN ISO 14155;
* Patients with a known coagulopathy (congenital);
* Concurrent participation in another experimental intervention or drug study
* Unwilling or unable to provide informed consent.
* A patient whose Glasgow-Blatchford score is 1 or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Effective coagulation of of actual or potential non-variceal bleeding in the upper Gastrointestinal (GI) tract. | Perioperative
  Primary haemostasis at day 0 using microwave coagulation of active bleeding or pre-coagulation of exposed vessels.

SECONDARY OUTCOMES:
Identification and incidence of intra-procedural complications | Day 0
Identification and incidence of post-procedural complications | At 24-72 hours, 1 week and 4 weeks
Change in Glasgow-Blatchford score | Day 0 for initial screen and then 24-72 hours post-procedure for second score.
  The Glasgow-Blatchford score will be recorded prior to and after microwave intervention

OTHER OUTCOMES:
Questionnaire assessment of device injection features | Perioperative
  Endoscopist assessment of injection functionality (questionnaire)
Questionnaire assessment of device adhesion characteristics | Perioperative
  Endoscopist assessment of tissue sticking (questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- East Kent Hospitals University Nhs Foundation Trust, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No